CLINICAL TRIAL: NCT03662893
Title: Checklist to Increase Effectiveness of Behavioural Therapy for Overactive Bladder
Brief Title: Behavioural Therapy With Checklist for Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Collaborators: Ministry of Health, Turkey (Other Government)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5002
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; behavioural therapy; adherence; drug persistence
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Group I were instructed to apply only written guideline forms of behavioural therapy which were the same as those in the checklist, Group II were instructed to apply behavioural therapy with a written checklist for patients to fully complete and Group III received medical treatment plus behavioural therapy without checklist. Group IV received medical treatment with a written checklist to fully complete
Who Masked: Outcomes Assessor
Masking Description: Analysis of treatment response was performed by a single independent urologist blinded to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Behavioural therapy with written guideline (Sham Comparator): Patients were instructed to apply only written guideline forms of behavioural therapy which were the same as those in the checklist over six-month period.
  Interventions: Behavioral: behavioural therapy with written guideline
- Behavioural therapy with checklist (Active Comparator): Patients were instructed to apply behavioural therapy with a written checklist for patients to fully complete over six-month period.
  Interventions: Behavioral: behavioural therapy with written checklist form to complete
- antimuscarinic drug plus verbal behavioural therapy (Active Comparator): Patients received medical treatment (once or twice per day) plus behavioural therapy without checklist over six-month period.
  Interventions: Drug: Antimuscarinic drugs used in overactive bladder; Behavioral: behavioural therapy with written guideline
- antimuscarinics plus checklist (Active Comparator): Patients received medical treatment (once or twice per day) with a written checklist to fully complete over six-month period.
  Interventions: Behavioral: behavioural therapy with written checklist form to complete; Drug: Antimuscarinic drugs used in overactive bladder

INTERVENTIONS:
Behavioral: behavioural therapy with written checklist form to complete — Behavioural therapy for overactive bladder such as advice on fluid balance, bladder retraining, urgency suppression or normal voiding techniques, pelvic floor muscle training, caffeine reduction, dietary changes, weight loss and other life style changes
  Arms: Behavioural therapy with checklist; antimuscarinics plus checklist
Drug: Antimuscarinic drugs used in overactive bladder — Antimuscarinic drugs (Tolterodine, solifenacin, propiverine, darifenacin,fesoterodine)
  Arms: antimuscarinic drug plus verbal behavioural therapy; antimuscarinics plus checklist
Behavioral: behavioural therapy with written guideline — behavioural therapy with written guideline,which are the same as those in the checklist
  Arms: Behavioural therapy with written guideline; antimuscarinic drug plus verbal behavioural therapy

SUMMARY:
The aim of this study is to investigate the efficiency of this newly-established checklist for overactive bladder (OAB) and whether determinate to adherence and persistence rate of combination of behavioural therapy and anticholinergic medications in patients with OAB.

DETAILED DESCRIPTION:
Overactive bladder (OAB) can worsen quality of life but it is not life-threatening condition. Although OAB medications effectively decrease disturbing symptoms of OAB, there are a lot of adverse side effects such as dry mouth, cognitive changes, constipation, urinary retention, blurred vision and dyspepsia. Therefore, guidelines have firstly recommended behavioural therapy which are noninvasive and not linked with adverse side effects. These behavioural recommendations include an advice on fluid balance, bladder retraining, urgency suppression or normal voiding techniques, pelvic floor muscle training, caffeine reduction, dietary changes, weight loss and other life style changes to improve lower urinary tract symptoms of OAB.

Educational leaflets, verbal or audio-visual instructions and trainings for behavioural therapy have been recommended for patients with OAB, however, to date these beneficial instructions have not been documented as a written checklist. Therefore, they were collected and developed as a written checklist to instruct the patients. The aim of this study was to investigate the efficiency of this newly-established checklist for OAB and whether determinate to adherence and persistence rate of combination of behavioural therapy and anticholinergic medications in patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

Patients with

* >8 micturitions,
* >1 nocturia,
* >6 urgency or
* >3 urgency urinary incontinence episodes per 24 h according to 3-day bladder diary.

Exclusion Criteria:

* active urinary tract infection,
* a maximum flow rate of 15 ml. per second or less at least 2 uroflow studies,
* residual volume of 100 cc or more,
* any medications for OAB, benign prostatic obstruction,
* polyuria (>3 l per 24 hour),
* endocrinological disease such as diabetes mellitus or diabetes insipidus which can cause polyuria,
* neurological or psychological disease disease,
* prostate or bladder cancer, renal disease, hypertension, genitourinary or congenital abnormality,
* history of transobturator or transvaginal tape or pelvic organ prolapse surgery
* pelvic radiation or surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Urinary frequency | 6 months
  >8 micturitions per day
Urgency | 6 months
  >6 urgency episodes per day

SECONDARY OUTCOMES:
Treatment Benefit Scale | 6 months
  Treatment Benefit Scale is consisted of four category including a score of 1 (greatly improved) or 2 (improved) is considered ''yes,'' and a score of 3 (not changed)or 4 (worsened) was considered ''no''
Urgency urinary incontinence | 6 months
  >3 urgency urinary incontinence episodes per day
Nocturia | 6 months
  >1 micturition at night

CONTACTS AND LOCATIONS:
Overall Officials: Koray Agras, Prof, Study Chair — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dumoulin C, Hunter KF, Moore K, Bradley CS, Burgio KL, Hagen S, Imamura M, Thakar R, Williams K, Chambers T. Conservative management for female urinary incontinence and pelvic organ prolapse review 2013: Summary of the 5th International Consultation on Incontinence. Neurourol Urodyn. 2016 Jan;35(1):15-20. doi: 10.1002/nau.22677. Epub 2014 Nov 15. PMID 25400065
- [Result] Gezginci E, Iyigun E, Yilmaz S. Comparison of 3 Different Teaching Methods for a Behavioral Therapy Program for Female Overactive Bladder: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2018 Jan/Feb;45(1):68-74. doi: 10.1097/WON.0000000000000398. PMID 29300292